CLINICAL TRIAL: NCT06205459
Title: Deep Marginal Acquisition With Thermacut Bur Versus Functional Crown Lengthening in Management of Deep Subgingival Interproximal Carious Lesions: A One Year Follow-up Randomized Controlled Trial
Brief Title: Deep Marginal Acquisition With Thermacut Bur Vs. Functional Crown Lengthening in Deep Carious Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Khairy Elmorsy, Master degree candidate, Conservative dentistry department, faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: thermacut bur dentsply
Record Dates: First submitted 2020-04-26; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Deep Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): deep marginal acquisition using thermacut bur from dentsply
  Interventions: Procedure: deep marginal acquisition using thermacut bur
- control (Active Comparator): functional crown lengthening
  Interventions: Procedure: deep marginal acquisition using thermacut bur

INTERVENTIONS:
Procedure: deep marginal acquisition using thermacut bur — thermacut bur is a tool which doesn't contain any abrasives so it is much safer on the root surface of both prepared and adjacent teeth, and yields better treatment outcome in cases when exposing deep margins is needed.
  Other Names: thermacut bur from dentsply

SUMMARY:
this clinical trial is conducted to compare between deep marginal acquistion by the means of thermacut bur Vs. functional crown lengthening in exposing deep subgingival interproximal cervical lesions

DETAILED DESCRIPTION:
Deep subgingival margins pose a great difficulty during restorative work with composite restorations. Exposing cavity margins is paramount in order to attain proper isolation, matrix adaptation and composite placement.

Several methods have been proposed to overcome the problem of exposing deep margins; functional crown lengthening is considered the gold standard of care regarding exposure of deep margins.

However, functional crown lengthening can pose many problems including the risk of root exposure, furcation involvement and compromising crown root ratio, besides risk of thread exposure if it is done beside implant, removal of bone from adjacent teeth and from buccal and lingual walls in order to create smooth bone architecture, and the complications of surgery such as post-operative pain, inflammation and edema and the risk of excessive bleeding.

Deep marginal acquisition and deep marginal extension (DMA & DME) are considered as a viable option in treating deep subgingival extended margins.

Several methods regarding deep marginal acquisition have been proposed including the use of diode laser and Electrosurgery, there is another protocol for exposing the gingival seat by the use of thermacut bur.

The rationale behind conducting this research is to propose an easy and predictable way to expose deep subgingival margins, without the need to perform surgical intervention.

The technique is done by clinicians with good outcomes, but never been tested or validated, this study is performed to verify whether this test should be validated or not.

ELIGIBILITY:
Inclusion Criteria:

- Subject not less than 18 years of age

1. Males or females
2. Community-dwelling
3. Have at least one deep subgingival interproximal carious lesion.
4. Can comply to oral hygiene measures or with good oral hygiene
5. Have sufficient cognitive ability to

5- Understand consent procedures.

Exclusion Criteria:

1. Patients less than 18 years old.
2. Disabilities:
3. Systemic diseases or severe medically compromised. (Cardiovascular disorder, diabetes, hypertensive, epileptic).
4. Lack of compliance.
5. Gingival hyperplasia, blood disorder.
6. Cognitive impairment.
7. Attachment loss signs of periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-02 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction: visual analogue scale | immediate post operative, 3 month, 6 month and 1 year
  using visual analogue scale

SECONDARY OUTCOMES:
Pocket depth and biological width | immediate post operative, 3 month, 6 month and 1 year
  Graded Periodontal Probe and (digital radiograph) bitewing with paralleling technique

OTHER OUTCOMES:
marginal integrity | immediate post operative, 3 month, 6 month and 1 year
  using modified USPHS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Cairo university, Cairo, Egypt